CLINICAL TRIAL: NCT02018068
Title: Postoperative Patient-controlled Perineural Analgesia After Orthopedic Surgery: A Medico-economic Comparative Evaluation of Patient Management by Remote Control Versus Bedside Care
Brief Title: Postoperative Patient-controlled Perineural Analgesia After Orthopedic Surgery by "Remote Control" Versus "Bedside Care"
Acronym: MICREL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9202
Record Dates: First submitted 2013-12-10; First posted 2013-12-23 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Injury of Foot, Shoulder or Knee; Perineural Analgesia; Pain, Postoperative
Keywords: Patient-controlled Perineural analgesia; Postoperative; Orthopedic surgery; "Remote Control" versus "at bedside care"; Comparative medico-economic evaluation
MeSH Terms: conditions — Foot Injuries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote control (Experimental): For patient randomized in arm "Remote Control", the communication with anesthesiologist will be done by teletransmission. The intervention "Remote control" is assigned to this arm. When evaluated pain values, sensory or motricity blockades are over the selected threshold then, the patient enters the data in the PCA (Patient Control Analgesia) pump, the physician in charge of the patient for the protocol is alerted by SMS on a specific smart phone and makes the necessary settings changes by Remote Control on the Micrel CareTM site.
  Interventions: Other: Remote control
- At bedside care (Active Comparator): For patient randomized in arm "At bedside care", the communication with the anesthesiologist in charge of the patient will be done via the nurses and referent physician of the medical unit, as a routine procedures. The necessary changes of pump settings are doing by the anesthesiologist. The intervention "at beside care" is assigned to arm "at bedside care".
  Interventions: Other: At bedside care

INTERVENTIONS:
Other: Remote control — When pain or sensory and motor block evaluation exceed the thresholds, the patient enters the data in the PCA (patient Control Analgesia) pump. The investigator is alerted by SMS on his smartphone and makes the necessary programming changes by remote control on the Micrel Care TM site. Systematic assessments via the PCA pump are scheduled for 9:00, 13:00 and 19:00 every day during 48 to 72 hours. The patient can alert his physician through his PCA pump of any additional requests (pain, motor blockade, numbness). The anesthesiologist receives an SMS alert and can make any necessary programming changes to the pump via the remote control.
  Arms: Remote control
Other: At bedside care — When pain or sensory and motor block evaluation exceed the thresholds, the nurse contacts the physician and she will be able to modify the pump settings according to the anesthesiologist prescription. The delay between the call of the patient and the programming changes, the duration of the procedure are reported. Systematic evaluations via the PCA (Patient Control Analgesia) pump are done when the patient arrives in this surgical ward and at 9:00, 13:00 and 19:00 every day for 48 to 72 hours.Throughout the study, if necessary, the nurse or referring physician performs the programming changes directly on the PCA pump and notes the delay in treatment. All the reasons and the duration of any bedside visit are reported.
  Arms: At bedside care

SUMMARY:
Perineural injection of local anesthesic is currently the reference method for the treatment of post operative pain in a patient undergoing major orthopedic surgery. Postoperative pain is a dynamic phenomena in every patient. It is classified as intense during the first postoperative hours after surgery, and decreases in a non-linear manner over the days following the procedure. PCA (patient control analgesia) infusion of local anesthesic allows an adaptation of the local analgesia doses to the evaluated pain scores, as well as permit a decrease in adverse events related to the continuous infusion technique (motor or sensory blockade, paresthesia, etc.). The physician can also modify the pump settings according to the postoperative rehabilitation plan.The use of new communication techniques such as "telemedecine" may be of interest in reducing treatment onset time and optimizing pain management. The remote control consists to change the settings of the pump after if the anesthesiologist was informed in real time (via a smartphone or a tablet) on patient pain level, sensory and motor blockades. The physician goes to a dedicated website (Micrel CareTM). and makes the necessary changes by remote control via a GPRS (General Packet Radio Service) connexion. The aim of this prospective, comparative, multicentric trial is to compare the effectiveness of patient management through two communication modalities: remote control versus bedside care.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective orthopedic surgery
* Patients older than 18 years old
* Patient with a surgical indication (foot, shoulder or knee) which can require placement of a perineural catheter
* Patients classified ASA class I to III
* Informed consent

Exclusion Criteria:

* Contraindication to regional anesthesia or local anesthetics
* Contraindication to paracetamol, ketoprofen or morphine (depending on the selected rescue analgesia)
* Hospital discharge less than 48 hours after surgery
* Psychomotor disease (teletransmission contraindication)
* Patient undergoing surgery with a duration greater than 4 hours
* Patient with a duration of perineural catheter less than 48 hours
* Protected patient
* Patient enrolled in another study
* Patient who can't understand local language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Time between the patient's call and the change in Patient Control Analgesia (PCA) pump settings | from arriving at the ward after surgery until 72 postoperative hours

SECONDARY OUTCOMES:
Number of nursing interventions | from arriving at the ward after surgery until 72 postoperative hours
Duration of nursing interventions | from arriving at the ward after surgery until 72 postoperative hours
Post operative pain measured by VAS (Visual Analog Scale) | from before implementation of PCA until 72 postoperative hours
Amount of rescue analgesia | from implementation of PCA (Patient Control Analgesia) until 72 postoperative hours
Patient satisfaction Score at catheter removal (at 72 postoperative hours) | at 72 postoperative hours
Time until the start of physical therapy | from surgery until 72 postoperative hours
the physiotherapist's satisfaction scores | at 72 postoperative hours
Healthcare staff (nurse and physician) satisfaction scores | at 72 postoperative hours
Duration of hospital stay | At the end of hospital stay (an expected average of 72 postoperative hours)
Overall cost of patient management strategy | until end of postoperative patient management (an average of 72 postoperative hours)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier XC CAPDEVILA, MD, PhD, Principal Investigator — CHU Montpellier - Department of Anesthesiology and critical care, Lapeyronie University Hospital
Locations (4):
- France (2):
  - Department of Anesthesiology and critical care, Lapeyronie University Hospital, Montpellier
  - Anesthesia Réanimation Department, Hôpital Saint Roch, Nice
- A Schweitzer Hospital, Dordrecht, Netherlands
- Rachid Hospital, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Capdevila X, Macaire P, Bernard N, Biboulet P, Cuvillon P, Choquet O, Bringuier S. Remote transmission monitoring for postoperative perineural analgesia after major orthopedic surgery: A multicenter, randomized, parallel-group, controlled trial. J Clin Anesth. 2022 May;77:110618. doi: 10.1016/j.jclinane.2021.110618. Epub 2021 Dec 1. PMID 34863052